CLINICAL TRIAL: NCT04364854
Title: Speech Entrainment for Aphasia Recovery
Acronym: SpARc
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00091924; U01DC017521-01A1 (NIH)
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Aphasia; Aphasia Non Fluent; Stroke
Keywords: Aphasia; Speech Language Pathology; Therapy
MeSH Terms: conditions — Aphasia; Aphasia, Broca; Stroke | interventions — SET protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SET (Speech Entrainment Therapy) 3 weeks (Experimental)
  Interventions: Behavioral: SET (Speech Entrainment Therapy) 3 weeks
- SET (Speech Entrainment Therapy) 4.5 weeks (Experimental)
  Interventions: Behavioral: SET (Speech Entrainment Therapy) 4.5 weeks
- SET (Speech Entrainment Therapy) 6 weeks (Experimental)
  Interventions: Behavioral: SET (Speech Entrainment Therapy) 6 weeks
- No Therapy 6 weeks (Other)
  Interventions: Other: No Therapy 6 Weeks

INTERVENTIONS:
Behavioral: SET (Speech Entrainment Therapy) 3 weeks — 3 weeks of SET which consists of practicing fluent speech in real time with an audio-visual computer program
  Arms: SET (Speech Entrainment Therapy) 3 weeks
Behavioral: SET (Speech Entrainment Therapy) 4.5 weeks — 4.5 weeks of SET which consists of practicing fluent speech in real time with an audio-visual computer program
  Arms: SET (Speech Entrainment Therapy) 4.5 weeks
Behavioral: SET (Speech Entrainment Therapy) 6 weeks — 6 weeks of SET which consists of practicing fluent speech in real time with an audio-visual computer program
  Arms: SET (Speech Entrainment Therapy) 6 weeks
Other: No Therapy 6 Weeks — Participants will not be getting any SET for 6 weeks
  Arms: No Therapy 6 weeks

SUMMARY:
After a stroke, many people experience a language impairment called aphasia. One of the most debilitating types of aphasia is non-fluent aphasia. Non-fluent aphasia is defined by significantly reduced speech production, with the speaker producing only a few words or even less. Speech entrainment therapy (SET) is a treatment that has been shown to increase fluency in people with non-fluent aphasia. The study looks to define the best dose of SET that leads to sustained improvements in spontaneous speech production.

Participants who are eligible will undergo baseline language testing, an MRI, and will be randomized into one of 4 treatment groups: SET for 3 weeks, SET for 4.5 weeks, SET for 6 weeks, and no treatment (control group).

ELIGIBILITY:
Inclusion Criteria

* Aphasia as a result of a left hemisphere ischemic or hemorrhagic stroke (WAB-R Aphasia Quotient <93.8).
* Presence of left hemisphere stroke in clinical imaging (CT/MRI) and NIHSS
* Participants must have spoken English as their primary language.
* 21-81 years old
* Pre-stroke modified Rankin Scale (mRS)= 2 or less
* Post-stroke mRS= 4 or less.
* At least 6 months post-stroke.
* Non-fluent aphasia (WAB-R Comprehension score >4 and WAB-R Fluency score <6).
* Technological compatibility (to be determined by clinical judgment of SLP)

Exclusion Criteria

* History of chronic neurological or psychiatric diseases (excluding migraines, depression, or post-stroke epilepsy). Self-reported history of learning disability.
* Severe dysarthria (determined via SLP clinical judgment from spontaneous speech tasks on the ASRS 3.0).
* Global aphasia.
* History of right-hemisphere strokes or brain stem/cerebellar strokes with persistent deficits (as evidenced by MRI/CT and NIHSS).
* Uncorrectable hearing as determined by the SLP's clinical judgment.
* Uncorrectable vision.
* Contraindications to MRI or inability to complete the MRI scanning session.
* Women who are pregnant.

Ages: 21 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Bonilha, MD, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SET (Speech Entrainment Therapy) 3 weeks | SET (Speech Entrainment Therapy) 4.5 weeks | SET (Speech Entrainment Therapy) 6 weeks | No Therapy 6 weeks
Started | 20 | 20 | 20 | 20
Completed | 18 | 20 | 19 | 16
Not Completed | 2 | 0 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 3
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SET (Speech Entrainment Therapy) 3 Weeks | SET (Speech Entrainment Therapy) 4.5 Weeks | SET (Speech Entrainment Therapy) 6 Weeks | No Therapy 6 Weeks | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at the time of enrollment.
  years | 60.8 (11.6) | 56.8 (12.1) | 56.8 (15) | 57.4 (14.1) | 58 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 3 | 8 | 25
  Male | 13 | 13 | 17 | 12 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 20 | 19 | 19 | 76
  Unknown or Not Reported | 2 | 0 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 4 | 12
  White | 18 | 16 | 16 | 16 | 66
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Stroke Onset Age [Mean (Standard Deviation); unit: years] — Age of the participant at the time of stroke that resulted in chronic aphasia. Population: Participants that had available data.
  years
    number analyzed (Participants) | 19 | 20 | 20 | 20 | 79
    (all) | 55.1 (13.4) | 51.6 (14) | 52.6 (13.3) | 55.1 (15.4) | 53.5 (13.8)
VPM - Narrative [Mean (Standard Deviation); unit: verbs per minute] — Verbs per minute (VPM) will be assessed through narrative storytelling tasks - with four different stories. The narrative stories will be: 1) Cinderella story, 2) Little Red Riding Hood, 3) The Three Little Pigs, and 4) Goldilocks. Population: Participants with available data.
  verbs per minute
    number analyzed (Participants) | 20 | 19 | 20 | 17 | 76
    (all) | 8.7 (7.7) | 9.1 (11.5) | 3.1 (3.4) | 3.8 (3.7) | 6.2 (7.8)
VPM - Procedural [Mean (Standard Deviation); unit: verbs per minute] — Verbs per minute (VPM) will be assessed through procedural storytelling - with four different stories. The procedural stories are: 1) how to make a peanut butter and jelly sandwich, 2) how to make scrambled eggs, 3) how to brew coffee, and 4) how to wash dishes. Population: Participants with available data.
  verbs per minute
    number analyzed (Participants) | 20 | 20 | 19 | 17 | 76
    (all) | 5.8 (5.2) | 8.2 (8.6) | 4.7 (5.2) | 5.7 (5.3) | 6.1 (6.3)
VPM - Average [Mean (Standard Deviation); unit: verbs per minute] — Verbs per minute (VPM) will be assessed through procedural storytelling and narrative storytelling tasks - with four items in each category. The procedural storytelling items are: 1) how to make a peanut butter and jelly sandwich, 2) how to make scrambled eggs, 3) how to brew coffee, and 4) how to wash dishes.
  The narrative items will be: 1) Cinderella story, 2) Little Red Riding Hood, 3) The Three Little Pigs, and 4) Goldilocks.
  VPM is averaged between the procedural storytelling and narrative storytelling tasks. Population: Participants with available data.
  verbs per minute
    number analyzed (Participants) | 20 | 20 | 20 | 17 | 77
    (all) | 7.3 (5.8) | 8.5 (9.7) | 3.8 (3.1) | 4.8 (3.6) | 6.1 (6.4)
Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) [Mean (Standard Deviation); unit: score on a scale] — Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) is a health-related quality of life measure that evaluates a participant's physical, psychosocial, and communication functioning. The final score is a decimal number between 0 and 5 with 5 indicating the best quality of life. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 20 | 20 | 18 | 78
    (all) | 3.61 (0.67) | 3.59 (0.63) | 3.12 (0.67) | 3.43 (0.83) | 3.44 (0.72)
WAB-R [Median (Inter-Quartile Range); unit: score on a scale] — Western Aphasia Battery-Revised (WAB-R) is a common clinical aphasia assessment used to determine the presence of non-fluent aphasia. The final score (known as the aphasia quotient) takes a value between 0 to 100 with lower scores indicating more severe aphasia and higher scores indicating less severe aphasia.
  score on a scale | 43.5 [28.9 to 70.7] | 49.4 [33.5 to 69.4] | 46.3 [32.6 to 63.9] | 53.9 [25.8 to 70.6] | 47.8 [30 to 68.5]
ASRS [Median (Inter-Quartile Range); unit: score on a scale] — Apraxia of Speech Rating Scale (ASRS) assesses the apraxia of speech of participants. The final score takes a value between 0 and 52 with a lower score indicating less severe apraxia and higher scores indicating more severe apraxia. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 18 | 17 | 19 | 74
    (all) | 20 [9.5 to 26] | 18.5 [7 to 20] | 23 [18 to 25] | 17 [11 to 23] | 19 [11 to 23]
WAIS III Matrix Reasoning Raw Score [Median (Inter-Quartile Range); unit: score on a scale] — Wechsler Adult Intelligence Scale (WAIS) III is an overall assessment of intellectual abilities. Only the matrix reasoning subtest score will be reported here which assesses nonverbal reasoning abilities. This score takes a value between 0 and 26 with a higher score indicating better abilities. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 20 | 20 | 18 | 78
    (all) | 8 [5 to 13] | 12.5 [9 to 14] | 11.5 [7.5 to 14.5] | 13 [7 to 15] | 12 [7 to 14]
LOFT Score [Median (Inter-Quartile Range); unit: score on a scale] — Lexical Orthography Familiarity Test (LOFT) is a type of assessment used to measure how familiar someone is with the written forms of words. The score takes a value between 0 and 50 with a higher score indicating more familiarity with words. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 20 | 20 | 18 | 78
    (all) | 43.5 [33.5 to 49] | 44 [39.5 to 47.5] | 45 [40 to 49] | 49 [43 to 50] | 45.5 [38 to 49]
Pyramids and Palm Trees Test Score [Median (Inter-Quartile Range); unit: score on a scale] — The Pyramids and Palm Trees Test assesses a participant's ability to access semantic memory by identifying conceptual relationships between words and pictures. The score takes a value between 0 and 52 with a higher score indicating better semantic memory abilities. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 20 | 20 | 18 | 78
    (all) | 45.5 [38.5 to 49] | 45.5 [42.5 to 48] | 44 [42 to 47] | 47 [41 to 49] | 45.5 [41 to 48]
Post-Stroke Fatigue Score [Median (Inter-Quartile Range); unit: score on a scale] — The Vertical Numerical Rating Scale-Face Rating Scale is a measure of fatigue severity in a stroke patient. The score takes a value between 0 and 10 with 0 representing no fatigue and 10 representing extreme fatigue. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 20 | 20 | 18 | 78
    (all) | 2 [0 to 4] | 2 [0 to 4] | 3 [1.5 to 5.5] | 4 [2 to 5] | 2 [1 to 5]
RHHI-S Score [Median (Inter-Quartile Range); unit: score on a scale] — The Revised Hearing Handicap Inventory Screening (RHHIS) assesses the level of a participant's self-reported hearing difficulty. The score ranges from 0 to 40 with a higher score indicating more difficult hearing ability.
  score on a scale | 0 [0 to 8] | 0 [0 to 0] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 2]
Modified - PNT Score [Median (Inter-Quartile Range); unit: score on a scale] — The modified Philadelphia Naming Test (PNT) is a picture naming test that assesses word retrieval. The final score ranges from 0 to 175 with higher scores indicating better naming ability. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 20 | 20 | 18 | 78
    (all) | 18 [1 to 111] | 47 [8.5 to 109] | 25 [4.5 to 73.5] | 27 [0 to 83] | 32.5 [2 to 102]
Modified - PRT Score [Median (Inter-Quartile Range); unit: score on a scale] — The modified Philadelphia Repetition Test (PRT) assesses a participant's ability to orally repeat a name he/she heard. The score takes a value between 0 and 175 with a higher score indicating better repetition ability. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 20 | 20 | 18 | 78
    (all) | 92.5 [40 to 144] | 133 [74 to 157] | 94.5 [22.5 to 129.5] | 97.5 [26 to 146] | 102 [40 to 146]
SADQ Score [Median (Inter-Quartile Range); unit: score on a scale] — The Stroke Aphasia Depression Questionnaire (SADQ) is a measure of depression for people who have aphasia due to stroke. The final score ranges between 0 and 30 with higher scores indicating more severe depression. Population: Participants with available data.
  score on a scale
    number analyzed (Participants) | 20 | 20 | 20 | 18 | 78
    (all) | 10.5 [6.5 to 12.5] | 11 [8.5 to 14.5] | 9 [7.5 to 14] | 10 [7 to 14] | 10 [7 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Average Verbs Per Minute (VPM) Change From Baseline
Description: VPM will be assessed through procedural storytelling and narrative storytelling tasks - with four items in each category. The procedural storytelling items are: 1) how to make a peanut butter and jelly sandwich, 2) how to make scrambled eggs, 3) how to brew coffee, and 4) how to wash dishes.
  The narrative items will be: 1) Cinderella story, 2) Little Red Riding Hood, 3) The Three Little Pigs, and 4) Goldilocks.
  VPM is averaged between the procedural storytelling and narrative storytelling tasks.
Time Frame: 3 months after treatment (or no treatment)
Population: Participants with available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: verbs per minute
Arm/Group | SET (Speech Entrainment Therapy) 3 weeks | SET (Speech Entrainment Therapy) 4.5 weeks | SET (Speech Entrainment Therapy) 6 weeks | No Therapy 6 weeks
Number analyzed (Participants) | 20 | 20 | 20 | 18
verbs per minute | 0.3 [-1.25 to 1.86] | 0.62 [-2.15 to 3.39] | -0.26 [-1.96 to 1.43] | 0.52 [-0.85 to 1.89]
Statistical Analysis 1: Comparison: SET (Speech Entrainment Therapy) 3 weeks vs No Therapy 6 weeks; Test type: Other — This study was not designed to perform a hypothesis test. No p-values will be reported; Mean Difference (Net) = -0.22, 95% CI 2-sided [-2.31 to 1.87] — Analyzed using a repeated measures model that included the following fixed affects: categorical visit by treatment group interaction, site, baseline aphasia severity score, baseline VPM, and age
Statistical Analysis 2: Comparison: SET (Speech Entrainment Therapy) 4.5 weeks vs No Therapy 6 weeks; Test type: Other — This study was not designed to perform a hypothesis test. No p-values will be reported; Mean Difference (Net) = 0.1, 95% CI 2-sided [-2.94 to 3.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: SET (Speech Entrainment Therapy) 6 weeks vs No Therapy 6 weeks; Test type: Other — This study was not designed to perform a hypothesis test. No p-values will be reported; Mean Difference (Net) = -0.78, 95% CI 2-sided [-2.9 to 1.33] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) Change From Baseline
Description: Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) is a health-related quality of life measure that evaluates a participant's physical, psychosocial, and communication functioning. The final score is a decimal number between 0 and 5 with 5 indicating the best quality of life.
Time Frame: 3 months after treatment (or no treatment)
Population: Participants that have available data and did not withdraw consent prior to completing the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SET (Speech Entrainment Therapy) 3 weeks | SET (Speech Entrainment Therapy) 4.5 weeks | SET (Speech Entrainment Therapy) 6 weeks | No Therapy 6 weeks
Number analyzed (Participants) | 20 | 20 | 20 | 18
score on a scale | 0 [-0.15 to 0.15] | 0.1 [-0.11 to 0.3] | -0.16 [-0.3 to -0.02] | 0.06 [-0.06 to 0.19]
Statistical Analysis 1: Comparison: SET (Speech Entrainment Therapy) 3 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.26 to 0.13] — Analyzed using a repeated measures model that included the following fixed affects: categorical visit by treatment group interaction, site, baseline aphasia severity score, baseline SAQOL-39, and age
Statistical Analysis 2: Comparison: SET (Speech Entrainment Therapy) 4.5 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.21 to 0.28] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: SET (Speech Entrainment Therapy) 6 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.42 to -0.04] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Narrative Verbs Per Minute (VPM)
Description: VPM will be assessed through narrative storytelling tasks - with four different stories. The narrative stories will be: 1) Cinderella story, 2) Little Red Riding Hood, 3) The Three Little Pigs, and 4) Goldilocks.
Time Frame: 3 months after treatment (or no treatment)
Population: Participants that have available data and did not withdraw consent prior to completing the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: verbs per minute
Arm/Group | SET (Speech Entrainment Therapy) 3 weeks | SET (Speech Entrainment Therapy) 4.5 weeks | SET (Speech Entrainment Therapy) 6 weeks | No Therapy 6 weeks
Number analyzed (Participants) | 20 | 20 | 20 | 18
verbs per minute | 0.25 [-1.92 to 2.43] | 0.89 [-1.71 to 3.49] | 0.35 [-1.74 to 2.44] | 0.1 [-1.56 to 1.75]
Statistical Analysis 1: Comparison: SET (Speech Entrainment Therapy) 3 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = 0.16, 95% CI 2-sided [-2.59 to 2.9] — Analyzed using a repeated measures model that included the following fixed affects: categorical visit by treatment group interaction, site, baseline aphasia severity score, baseline VPM - Narrative, and age
Statistical Analysis 2: Comparison: SET (Speech Entrainment Therapy) 4.5 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = 0.79, 95% CI 2-sided [-2.23 to 3.8] — Analyzed using a repeated measures model that included the following fixed affects: categorical visit by treatment group interaction, site, baseline aphasia severity score, baseline VPM-Narrative, and age
Statistical Analysis 3: Comparison: SET (Speech Entrainment Therapy) 6 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = 0.25, 95% CI 2-sided [-2.32 to 2.82] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Procedural Verbs Per Minute (VPM) Change From Baseline
Description: Verbs per minute (VPM) will be assessed through procedural storytelling - with four different stories. The procedural storytelling items are: 1) how to make a peanut butter and jelly sandwich, 2) how to make scrambled eggs, 3) how to brew coffee, and 4) how to wash dishes.
Time Frame: 3 months after treatment (or no treatment)
Population: Participants that have available data and did not withdraw consent prior to completing the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: verbs per minute
Arm/Group | SET (Speech Entrainment Therapy) 3 weeks | SET (Speech Entrainment Therapy) 4.5 weeks | SET (Speech Entrainment Therapy) 6 weeks | No Therapy 6 weeks
Number analyzed (Participants) | 20 | 20 | 20 | 18
verbs per minute | 0.77 [-1.78 to 3.31] | 1.1 [-2.58 to 4.79] | -1.27 [-4.2 to 1.67] | 0.84 [-1.65 to 3.33]
Statistical Analysis 1: Comparison: SET (Speech Entrainment Therapy) 3 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = -0.07, 95% CI 2-sided [-3.59 to 3.45] — Analyzed using a repeated measures model that included the following fixed affects: categorical visit by treatment group interaction, site, baseline aphasia severity score, baseline VPM - Procedural, and age
Statistical Analysis 2: Comparison: SET (Speech Entrainment Therapy) 4.5 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = 0.27, 95% CI 2-sided [-4.27 to 4.8] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: SET (Speech Entrainment Therapy) 6 weeks vs No Therapy 6 weeks; Test type: Other — This trial was not designed for hypothesis testing. No p-values will be reported; Mean Difference (Net) = -2.11, 95% CI 2-sided [-5.77 to 1.56] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months after treatment (or no treatment).
Arm/Group | SET (Speech Entrainment Therapy) 3 weeks | SET (Speech Entrainment Therapy) 4.5 weeks | SET (Speech Entrainment Therapy) 6 weeks | No Therapy 6 weeks
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/20 | 2/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SET (Speech Entrainment Therapy) 3 weeks (N=20) | SET (Speech Entrainment Therapy) 4.5 weeks (N=20) | SET (Speech Entrainment Therapy) 6 weeks (N=20) | No Therapy 6 weeks (N=20)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post stroke seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SET (Speech Entrainment Therapy) 3 weeks (N=20) | SET (Speech Entrainment Therapy) 4.5 weeks (N=20) | SET (Speech Entrainment Therapy) 6 weeks (N=20) | No Therapy 6 weeks (N=20)
Anxiety (Psychiatric disorders) | NA | NA | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT04364854/Prot_001.pdf
  • Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04364854/SAP_002.pdf
  • Informed Consent Form (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT04364854/ICF_003.pdf